CLINICAL TRIAL: NCT07399470
Title: Randomized, Open-label, Single-dose, Crossover Study to Compare the Pharmacokinetics and Safety/Tolerability of a Triple Fixed-dose Combination Tablet (Gemigliptin/Dapagliflozin/Metformin) 50/10/1000 mg and Co-administered Zemiglo (Gemigliptin) 50 mg and Xigduo XR (Dapagliflozin/Metformin) 10/1000 mg in Healthy Adult Subjects Under Fasting Conditions
Brief Title: A Clinical Study in Healthy Adults to See How the Body Processes and How Safe a Tablet That Combines Gemigliptin, Dapagliflozin, and Metformin is, Compared With Taking Zemiglo and Xigduo XR Together While Fasting.
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: LG-GMCL003
Record Dates: First submitted 2026-01-23; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Healthy Volunteers; Fasting Conditions
Keywords: Fasting conditions; Healthy Volunteers; Bioequivalence Study
MeSH Terms: interventions — Drug Evaluation; dapagliflozin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): test drug > reference drug
  Interventions: Drug: Test drug: Fixed-dose combination of gemigliptin/dapagliflozin/metformin 50/10/1000 mg; Drug: Reference drug: Gemigliptin (Zemiglo) 50mg, Dapagliflozin/metformin (Xigduo XR) 10/1000 mg
- Sequence 2 (Experimental): reference drug > test drug
  Interventions: Drug: Test drug: Fixed-dose combination of gemigliptin/dapagliflozin/metformin 50/10/1000 mg; Drug: Reference drug: Gemigliptin (Zemiglo) 50mg, Dapagliflozin/metformin (Xigduo XR) 10/1000 mg

INTERVENTIONS:
Drug: Test drug: Fixed-dose combination of gemigliptin/dapagliflozin/metformin 50/10/1000 mg — All participants will take 1 tablet of either test drug or 2 tablets of reference drug with fasting conditions.
Drug: Reference drug: Gemigliptin (Zemiglo) 50mg, Dapagliflozin/metformin (Xigduo XR) 10/1000 mg — All participants will take 1 tablet of either test drug or 2 tablest of reference drug with fasting conditions.

SUMMARY:
Bioequivalence study for the fixed-dose combination of Gemigliptin/Dapagliflozin/Metformin 50/10/1000 mg under fasting conditions in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults between 19 and 50 years of age
* People with a body weight within a healthy range
* People who do not have serious medical conditions and have been generally healthy in recent years
* People whose screening tests (blood tests, urine tests, vital signs, ECG, etc.) show no significant abnormalities
* Women of childbearing potential must not be pregnant at screening
* Participants must agree to use reliable contraception or abstain from sexual activity during the study and for a short period after the last dose
* People who fully understand the study, agree to follow study requirements, and provide written informed consent

Exclusion Criteria:

* People with a history of significant diseases, such as heart, liver, kidney, lung, neurological, psychiatric, immune, or cancer-related conditions
* People with digestive diseases or surgeries that may affect how medicines are absorbed
* People with abnormal screening laboratory results, especially related to liver or kidney function
* People who drink large amounts of alcohol, use drugs, or smoke heavily
* People who have recently taken certain medications, herbal products, or dietary supplements that could interfere with the study
* People who have recently participated in another clinical trial, donated blood, or received a blood transfusion
* Pregnant or breastfeeding women
* People with unstable or serious health conditions that could increase risk or affect study results
* Anyone who, in the opinion of the study doctor, is not suitable to participate

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2026-01-09 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
The plasma concentration of Gemigliptin, Dapagliflozin and Metformin | Up to 72 hours
  Area under the plasma concentration versus time curve (AUClast) of Gemigliptin, Dapagliflozin, and Metformin
The plasma concentration of Gemigliptin, Dapagliflozin and Metformin | Up to 72 hours
  Peak Plasma Concentration (Cmax) of Gemigliptin, Dapagliflozin, and Metformin

SECONDARY OUTCOMES:
The plasma concentration of Gemigliptin, Dapagliflozin and Metformin. | Up to 72 hours
  Time to Maximum Concentration(Tmax) of Gemigliptin, Dapagliflozin, and Metformin
The plasma concentration of Gemigliptin, Dapagliflozin and Metformin | Up to 72 hours
  Lag Time(Tlag) of Gemigliptin, Dapagliflozin, and Metformin
The plasma concentration of Gemigliptin, Dapagliflozin and Metformin | Up to 72 hours
  Area Under the Curve to Infinity(AUCinf) of Gemigliptin, Dapagliflozin, and Metformin
The plasma concentration of Gemigliptin, Dapagliflozin and Metformin | Up to 72 hours
  Half-life(t1/2) of Gemigliptin, Dapagliflozin, and Metformin
The plasma concentration of Gemigliptin, Dapagliflozin and Metformin | Up to 72 hours
  Apparent Clearance(CL/F) of Gemigliptin, Dapagliflozin, and Metformin

CONTACTS AND LOCATIONS:
Overall Officials: Seol Ju Moon, M.D., Professor, Principal Investigator — Jeonbuk National University Hospital
Locations (1):
- Jeonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea

IPD SHARING:
Plan to Share IPD: No